CLINICAL TRIAL: NCT06809907
Title: Kintsugi Voice Device SCID-5 Pivotal Study
Brief Title: Kintsugi Voice Device Pivotal Study
Status: Recruiting | Type: Observational
Sponsor: Kintsugi Mindful Wellness, Inc. (Industry)
Collaborators: Kolby Walker, DO (Unknown); Sonar Strategies (Unknown); Brittany Kimble (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20245287
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Depression; Depression Moderate; Depression Severe; Depression Mild
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Kintsugi Voice Device — The Kintsugi Voice Device is intended to be used to screen for the presence of voice signals consistent with a current moderate to severe depressive episode in patients aged 22 and older. The device is intended to be used by care providers licensed to screen for depression and in settings where the screening for depression occurs. The device is neither to be used in lieu of a complete patient evaluation nor to supplant any of the clinician's standard assessments for the screening or diagnosis of depression. The Kintsugi Voice Device is comprised of a software API and machine learning model that utilizes recorded voice samples as inputs and outputs the detection of signals consistent with current moderate to severe depressive episode as outputs.

SUMMARY:
A prospective, single arm, non-randomized, pivotal clinical validation study to evaluate the ability of the Kintsugi Voice Device (the Device) to aid clinical assessment for depression by comparing its output with a diagnosis made by a clinician using the Structured Clinical Interview for DSM-5 (SCID-5-RV) for up to 1000 English speaking adult patients ages 22 and older living in the United States. Recruitment will occur for 1 year and participation will be for up to 2 weeks

ELIGIBILITY:
Inclusion Criteria:

Age >22 at the time of informed consent Self-reported disruption to activities of daily living (e.g. missed scheduled healthcare appointments, unable to concentrate on tasks like reading, working, or completing daily activities, or difficult completing activities such as exercise, diet, or recreation) Access to a laptop, smartphone, tablet, or other device with a functioning microphone and access to the Internet Stated willingness to be video and audio recorded as part of the study Stated willingness to comply with all study procedures and availability for the duration of the study Functional English capacity in the home environment Availability for the duration of the study Resides in the United States at the time of consent and during completion of study

-

Exclusion Criteria:

* Participants with at least one of the following conditions will be excluded:

Any impairment that impacts their ability to speak and/or use a computer to complete online surveys and/or a virtual clinician assessment (E.g., visual impairment, motor impairment, and/or hearing impairment) Any lifetime history of neurological disease that impacts their ability to speak and/or use a computer to complete online surveys and/or a virtual clinician assessment (E.g., Central Nervous System disorders, Multiple Sclerosis, Amyotrophic Lateral Sclerosis, and/or Parkinson's Disease) Any lifetime history of Stroke, cognitive defect (E.g., dementia or Alzheimer's disease), and/or Traumatic Brain Injury Presence of voice disorders that impacts their ability to speak (E.g., acute or chronic laryngitis, vocal cord paresis or paralysis, or spasmodic dysphonia) Past or active heavy smokers (an average of >20 cigarettes per day) Subjects who have previously participated in any Kintsugi-sponsored study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll up to 1000 English speaking subjects >22 years old. Only subjects who meet all eligibility criteria and sign the informed consent will be enrolled. Participants who do not meet the criteria required for participation will not be presented with the opportunity to participate. Screen failures will not be considered a part of this research study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
1. Sensitivity and Specificity of Kintsugi Voice Device Relative to the SCID-5 | Day 1
  Achieve a composite lower bound of sensitivity greater than or equal to 70% and specificity greater than or equal to 70% for the KV Device relative to the high diagnostic confidence clinical reference standard as defined in Section 7.4.1 for which the device provides a result

SECONDARY OUTCOMES:
Adjudicated Samples Sensitivity and Specificity | Day 1
  Evaluate sensitivity and specificity for all adjudicated samples for which the device provides a result
PPV and NPV Evaluation | Day 1
  Evaluate the Positive Predictive Value (PPV) and Negative Predictive Value (NPV)
Subgroup Analysis (Sensitivity and Specificity) | Day 1
  Perform subgroup analyses including but not limited to age, race, and ethnicity
Indeterminate Result Analysis | Day 1
  Measurement of the proportion of all participants for whom the device provides no result

CONTACTS AND LOCATIONS:
Locations (1):
- Kintsugi (Decentralized, Virtual Study), Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No